CLINICAL TRIAL: NCT05479019
Title: Human Perception on Medical Extended Reality Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: USFDA
Record Dates: First submitted 2022-07-18; First posted 2022-07-28 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive stimuli (Experimental): Images/trials that contain a target
  Interventions: Behavioral: Visual stimuli
- Negative stimuli (Experimental): Images/trials that do not contain a target
  Interventions: Behavioral: Visual stimuli

INTERVENTIONS:
Behavioral: Visual stimuli — Stimuli will be shown to participants and they will be asked to perform a visual task.

SUMMARY:
The proposed research will collect participant's responses that respond to questions about visibility of certain signals on an immersive mixed reality environment. These responses will be used to assess Head Mounted Display (HMD) quality and task performance. Other collected data may be included such as response time and eye movements.

Responses will be collected via an FDA application designed to work with a wide range of HMDs and able to display both 2D simple scenes and 3D complete scenes. This application allows a human observer to look at a signal (sinusoidal, disk, sphere, etc.) on a synthetic noisy background or a realistic 3D scene both in virtual reality and augmented reality immersive environments. The application will also provide instructions and a response interface for the observer to respond to questions related to the visibility and to gather task performance measurements.

Participants will not be asked to complete tasks that require specific training or skills. Any adult human with normal or corrected-to-normal vision that can wear an HMD is eligible to participate in this experiment.

Data collected will not include identifiable information. FDA will perform participant enrollment and data collection, ensuring management of PII in accordance with federal rule. Participants will be recruited at will and in person, using promotional materials only containing language within this document. Participants will sign the attached consent form either electronically or by hard copy.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 70 years old
* No gender requirement
* No sensory, proprioceptive, or neural impairments
* Ability to sit for 20-30 minutes at a time, for up to 2 hours with 5-10 minute breaks
* Adults with normal or corrected-to-normal vision that can wear an HMD comfortably.

  * For participants with corrected-to-normal vision and, in the case of an HMD that is not compatible with glasses, contact lenses will be required

Exclusion Criteria:

* History of light sensitivity, epilepsy, or seizures
* Uncorrected visual impairments
* Pregnant women
* Participants that have corrected-to-normal vision with glasses that cannot wear the HMD comfortably
* Presence of sensory, proprioceptive, neural, vestibular, or physical impairments that limit fine motor control, gross movement, normal ambulation, or ability to sit/stand as needed for the study
* Claustrophobia such that use of an HMD induces anxiety or other negative psychological response
* Cognitive impairments that limit the ability to comprehend simple written and verbal instructions or identify and locate objects in space
* Subjects with migraine headaches or that experience motion sickness
* Current or prior diagnosis of epilepsy, seizure disorder, dementia, migraines (especially with visual aura), or other neurological diseases
* Current medical condition predisposing to nausea, dizziness, or vertigo (e.g. Meniere's disease)
* Ongoing psychosis, hallucinations, or dissociative disorders affecting perception of reality
* Hypersensitivity to flashing light or motion
* Irritated skin or open wounds on the scalp and face where the AR/VR headset will rest
* Past history of use of hallucinogenic medications (e.g. LSD, mesclun, etc.)
* Prior cervical spine disorder or Brachial plexus disorder or shoulder joint disorder, or hand disorder or past surgery in any of the previous stated anatomic areas (as these might affect the use, responsiveness, and/or dexterity of upper extremities or hand-eye coordination)
* Subjects will be excluded from participation in this study if they answer yes to a screening question about taking various medications listed below: (n.b. the reasons for subject being excluded is also noted with the potential side-effects of the noted medication)

  * Antihistamines (e.g. diphenhydramine {Benadryl}, etc.) -- Drowsiness, dizziness, constipation, stomach upset, blurred vision, or dry mouth/nose/throat may occur.
  * Muscle relaxants (e.g. methocarbamol {Robaxin}, cyclobenzaprine {Flexeril}, carisoprodol {Soma} , etc.) -- Drowsiness, tiredness, clumsiness, headache, dizziness, lightheadedness, dry mouth, stomach upset, nausea/vomiting, or blurred vision may occur.
  * Analgesic medications (e.g. narcotics, Class II controlled substances such as propoxyphene {Darvon} , etc.) -- Low blood pressure, drowsiness, fainting, dizziness, nausea, vomiting, generalized weakness, a feeling of general discomfort called malaise.
  * Sleep medications (e.g. zolpridem {Ambien}, etc.) -- Daytime drowsiness, dizziness, weakness, feeling "drugged" or light-headed; tired feeling, loss of coordination; memory loss, stuffy nose, dry mouth, nose or throat irritation; nausea, constipation, diarrhea, upset stomach, headache, muscle pain, anxiety, depression, aggression, agitation, confusion, or hallucinations (hearing or seeing.) This is not a complete list of side effects and others may occur.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Display Human Perception Assessment | 2 years initially
  The experiment will test the Head Mounted Displays with visual tasks. These tasks will allow us to gather information about how different headsets show visual stimuli and how humans perceive them. We designed tasks that allow us to collect information about contrast, resolution, temporal artifacts, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- 10903 New Hampshire Ave, WO62, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
No IPD will be shared to other researchers unless required by the publication journal or other protocols.